CLINICAL TRIAL: NCT00624156
Title: Expressive Writing and Adjustment to Metastatic Breast Cancer
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Indiana University (Other)
Responsible Party: Sponsor
Other Study IDs: 08-011
Record Dates: First submitted 2008-02-15; First posted 2008-02-26 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1: emotional disclosure writing intervention
  Interventions: Behavioral: Writing Intervention
- 2: control writing
  Interventions: Behavioral: Writing Intervention

INTERVENTIONS:
Behavioral: Writing Intervention — Participants in the emotional disclosure condition will be instructed to write continuously for 20 minutes about their deepest thoughts and feelings regarding their cancer experience.
  Other Names: Over four sessions, I want you to write about your experience with cancer. In your writing, I; want you to really let go and explore your very deepest emotions and thoughts. It is critical that you; delve deeply.
  Groups: 1
Behavioral: Writing Intervention — Participants assigned to the control condition will be instructed to describe in a detailed, nonemotional manner their daily activities. The 20-minute writing task will be introduced as a time management intervention
  Other Names: Over four sessions, I want you to write about how you use your time. I am interested in; everything you do during the course of a day. I realize that you experience many emotions, but in; your writing I want you to focus only on the facts, not on your emotions.
  Groups: 2

SUMMARY:
We are doing this study to see if writing about life experiences helps women adjust to breast cancer that has spread. We will compare two groups. One group will write about their breast cancer experience. The other will write about their daily activities. What we learn from this study may help us to find new ways to help women cope with breast cancer that has spread.

ELIGIBILITY:
Inclusion Criteria:

* Women with Stage IV breast cancer
* Receiving cancer care at Memorial Sloan-Kettering Cancer Center
* At least 18 years of age
* Can speak, read, and write in English
* In the judgment of consenting professionals able to provide informed consent
* Score of 4 or higher on the distress thermometer (established cutoff score for probable distress; see Jacobsen et al., 2005)

Exclusion Criteria:

* Significant psychiatric or cognitive impairment (dementia/delirium, retardation, psychosis) that in the judgment of the investigators will preclude providing informed consent and participating in the intervention
* Currently engaging in expressive writing (e.g., journal writing that involves expressing one's feelings) on a daily basis
* Currently participating in intervention trials with similar endpoints • Male

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MSKCC clinics
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2008-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Determine the potential utility of expressive writing for enhancing existential well-being (i.e., increasing a sense of meaning and peace and reducing demoralization) among women with metastatic breast cancer. | conclusion of the study

SECONDARY OUTCOMES:
Determine the potential utility of expressive writing for reducing distress (i.e., depressive symptoms, anxiety, cancer-specific and general distress) among women with metastatic breast cancer. | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Katherine DuHamel, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Mosher CE, Duhamel KN, Lam J, Dickler M, Li Y, Massie MJ, Norton L. Randomised trial of expressive writing for distressed metastatic breast cancer patients. Psychol Health. 2012;27(1):88-100. doi: 10.1080/08870446.2010.551212. Epub 2011 Jul 8. PMID 21678181
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org